CLINICAL TRIAL: NCT04609280
Title: A Single-arm, Single-stage Phase II Trial of Selective Avoidance of Nodal VolumEs at Minimal Risk (SAVER) in the Contralateral Neck of Patients With p16-positive Oropharynx Cancer
Brief Title: Selective Avoidance of Nodal VolumEs at Minimal Risk (GCC 20110)
Acronym: SAVER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00093439
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Oropharynx Cancer; Oropharyngeal Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Oropharynx Cancer; Oropharyngeal Squamous Cell Carcinoma; Radiotherapy; Proton Therapy; Photon Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Reduced C/L elective nodal volume (Experimental): All patients will receive the reduced C/L elective nodal volume as described. Treatment will be delivered via IMRT/VMAT or PBPT.
  Interventions: Radiation: Intensity modulated radiotherapy (IMRT)/volumetric modulated arc therapy (VMAT) or Pencil beam proton therapy (PBPT)

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy (IMRT)/volumetric modulated arc therapy (VMAT) or Pencil beam proton therapy (PBPT) — Delivered over 6 weeks in 30 daily fractions in the adjuvant setting and over 6.5 weeks in 33 daily fractions in the definitive setting. In the adjuvant setting, areas with positive surgical margins or nodal stations with pathologic extranodal extension will receive 63 Gy. Margin negative resection bed and involved nodal stations without extranodal extension will receive 54 Gy. Low-risk elective nodal volumes (i.e. ceCTV) will receive 51 Gy. In the definitive setting, gross disease will receive 69.96 Gy, areas at high-risk for subclinical disease will receive 60 Gy, and areas at low-risk for harboring subclinical disease (i.e. ceCTV) will receive 52.8 Gy.

SUMMARY:
This is a phase II, non-randomized, therapeutic trial with the primary objective to determine the efficacy of reduced contralateral (C/L) elective nodal treatment volumes in preventing C/L recurrences at 2 years in patients with p16 positive oropharyngeal squamous cell carcinoma undergoing definitive or adjuvant RT.

DETAILED DESCRIPTION:
Patients with human papillomavirus (HPV) or its surrogate marker p16, positive oropharyngeal squamous cell carcinoma (p16+OPSCC) exhibit favorable overall survival (OS) rates of 70-100% at 3 years. These outcomes are dependent on disease burden and patient characteristics and independent of treatment modality. Significant treatment related side effects exist despite advances in radiotherapy (RT) technology, surgical techniques, and supportive care. In addition to common acute toxicities, the favorable OS of patients with p16+OPSCC potentially places them at increased risk for developing long-term treatment-induced side-effects. Therefore, it is important to establish novel management approaches that maintain excellent current clinical outcomes while effectively reducing acute and long-term side effects.

One such approach of limiting RT-induced toxicity is to decrease the amount of normal tissue that receives radiation through judicious reduction of RT treatment volumes. Treatment of elective nodal volumes increases dose to numerous organs at risk (OARs). Patients with well-lateralized tonsil tumors and limited neck disease can effectively be treated with ipsilateral nodal radiotherapy. However, based on recent phase III trials, contralateral (C/L) elective nodal radiation is performed for the majority of patients with p16+OPSCC increasing acute and long-term toxicities. Therefore, judicious data-driven approaches for decreasing the number of elective ipsilateral and contralateral nodal levels treated is necessary to limit RT-induced side effects. This protocol tests the hypothesis that treating only the high-risk sub-volumes of levels II and III would be effective in maintaining regional control in the elective neck while decreasing xerostomia (dry mouth) and dysphagia (swallowing difficulties).

ELIGIBILITY:
Inclusion Criteria:

1. Is there pathologically (histologically or cytologically) proven diagnosis of p16+ squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma) of the oropharynx (tonsil or base of tongue)? Note: Cytologic diagnosis from a cervical lymph node (from a paraffin block, not from smears) is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx. Clinical evidence should be documented, may consist of palpation, imaging, or endoscopic evaluation, and should be sufficient to estimate the size of the primary (for T stage).
2. Does the patient require elective contralateral radiotherapy in the definitive or adjuvant setting (i.e. base of tongue primary or tonsil with base of tongue invasion, soft palate invasion, or medialized as defined by > 1/3 of the distance from the tonsil to the midline of the soft palate?
3. Does the patient have clinical stage T1-4, N0, N1 or N3, and M0 disease (AJCC 8th edition) as defined by physical examination and appropriate imaging (PET/CT preferred, CT neck with IV contrast with CT chest without contrast as recommended alternative to PET/CT)?
4. Was a general history and physical examination performed by a radiation oncologist, medical oncologist, or head and neck surgeon within 60 days prior to registration?
5. Was the patient's Zubrod Performance Status 0-1 within 30 days prior to registration?
6. Is the patient ≥ 18 years of age?
7. For women of childbearing potential, was a serum pregnancy test completed within 2 weeks of initiation or radiotherapy?
8. If yes, was the serum pregnancy test negative?
9. If a woman of child-bearing potential or sexually active male, is the patient willing to use effective contraception throughout their participation in the treatment phase of the study and at least 180 days following the last study treatment.
10. Did the patient provide study specific informed consent prior to study entry, including consent for mandatory submission of tissue for required p16 review?

Exclusion Criteria:

1. Does the patient have cancer considered to be from an oral cavity site (oral tongue, floor mouth, alveolar ridge, buccal or lip), nasopharynx, hypopharynx, or larynx?
2. Does the patient have a carcinoma of the neck of unknown primary origin?
3. Does the patient have distant metastasis?
4. Does the patient have prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years?
5. Did the patient have prior systemic chemotherapy for the study cancer (prior chemotherapy for a different cancer is allowable)?
6. Did the patient have prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields?
7. Did the patient have prior surgery of the head and neck excluding superficial removal of cutaneous skin malignancies?
8. Is the patient homeless?
9. Does the patient have an active drug or alcohol dependency?
10. Is the patient pregnant or nursing (an exception will be made for nursing patients that are not receiving chemotherapy)?
11. Radiographic evidence of contralateral nodal disease as described below. 1) Max standardized uptake value (SUV) greater than 3.0, or 2) Short-axis diameter is > 1.5 cm for level II nodes, > 0.8 cm for retropharyngeal node, or > 1.0 cm for level III, IV, or V, or 3) Central necrosis or heterogeneous enhancement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Elective out-of-field contralateral nodal failure | 2-years following completion of radiotherapy
  Time to failure will be calculated from the date of informed consent until the date of nodal failure in the untreated elective neck sub-volume.

SECONDARY OUTCOMES:
Grade 2/3 xerostomia | 2-years following completion of radiotherapy
  defined by PRO-CTCAE (patient-reported outcome (PRO) measurement system - Common Terminology Criteria for Adverse Events (CTCAE))
Dysphagia using The M.D. Anderson Dysphagia Inventory (MDADI) | 2-years following completion of radiotherapy
  The M.D. Anderson Dysphagia Inventory is a self-administered questionnaire designed specifically for evaluating the impact of dysphagia on the Quality of Life (QOL) of patients with head and neck cancer.
PEG-tube rate | 2-years following completion of radiotherapy
  Percutaneous endoscopic gastrostomy (PEG)-tube rate
Overall survival | 2-years following completion of radiotherapy
Progression-free survival | 2-years following completion of radiotherapy
Locoregional control | 2-years following completion of radiotherapy
Incidence of pulmonary metastases | 2-years following completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Witek, MD, Principal Investigator — University of Maryland/Maryland Proton Treatment Center
Locations (6):
- United States (6):
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - UMMC, Baltimore, Maryland
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Upper Chesapeake Health, Bel Air, Maryland
  - Central Maryland Radiation Oncology, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No